CLINICAL TRIAL: NCT03395028
Title: Granulocyte-Colony Stimulating Factor Adjunct Therapy for Biliary Atresia
Brief Title: GCSF Adjunct Therapy for Biliary Atresia
Acronym: BA_GCSF
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Holterman, Ai-Xuan, M.D. (Individual)
Collaborators: T. Rose Clinical, Inc., United States (Unknown); Children's National Research Institute (Other); Big Leap Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CR00005169; IND 119679-0007 (Other: Food and Drug Administration)
Record Dates: First submitted 2017-12-22; First posted 2018-01-09 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Biliary Atresia
Keywords: Biliary Atresia; Granulocyte Colony Stimulating Factor; GCSF
MeSH Terms: conditions — Biliary Atresia | interventions — Granulocyte Colony-Stimulating Factor; Filgrastim

STUDY DESIGN:
Intervention Model Description: Dose determination for GCSF
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Granulocyte Colony-Stimulating Factor — G-CSF is a glycoprotein produced by monocytes, fibroblasts, and endothelial cells. Filgrastim is a human granulocyte colony stimulating factor (G-CSF) produced by recombinant DNA technology with NEUPOGEN® as the Amgen Inc. trademark for filgrastim. G-CSF regulates the production, proliferation and differentiation of neutrophils and hematopoietic stem cell precursors within the bone marrow leading to dose-dependent increase in circulating neutrophils and hematopoietic stem cells in the blood. It is indicated to reduce the incidence of infection in patients with severe neutropenia, for neutrophil recovery in neutropenic patients with bone marrow depletion, to mobilize hematopoietic progenitor stem cell for collection by leukapheresis in hematopoietic stem cell transplantation.
  Other Names: Filgrastim

SUMMARY:
The Investigators propose to test the hypothesis that GCSF therapy enhances the clinical outcome of Kasai operated Biliary Atresia (BA) patients. In this study, Investigators will conduct a dose determination for GCSF use in post Kasai subjects to support a future phase 2 efficacy study. The first 3 post Kasai BA subjects with liver biopsy-confirmed BA will be given 5 ug/kg/d of GCSF in 3 daily subcutaneous doses starting on post Kasai day 3. A second group of 3 subjects will be assigned to the 10 ug/Kg/d dose after the 5ug/kg/d dose has been proven to be safe. The levels of circulating hematopoietic stem cells and a 1-month safety profile will be analyzed.

DETAILED DESCRIPTION:
In BA, neonatal fibrous obliteration of the biliary tract obstructs biliary drainage and promotes biliary fibrosis. BA is the leading cause of pediatric chronic end-stage liver disease and pediatric liver transplantation. Relief of cholestasis by the Kasai portoenterostomy is only partly successful with continued progression of fibrosis to hepatic insufficiency and, for long term survival, with eventual need for liver transplantation in the majority of the patients. In animal models of liver injury, GCSF enhances hematopoietic stem cell HSC mobilization and engraftment in the liver with associated improved liver repair response and attenuated hepatic necrosis and fibrosis. Randomized controlled trials of GCSF intervention for chronic liver failure in adult patients with acute hepatic decompensation showed improved short-term survival and hepatic indices such the model for end-stage liver disease (MELD) scores.

The Investigators propose that post Kasai GCSF therapy attenuates biliary fibrosis and progression to cirrhosis. The objectives are meant to demonstrate that Kasai-GCSF sequential therapy improves biliary drainage, and delays the progression of hepatic insufficiency. Toward this goal, Investigators will first evaluate in post Kasai subjects the maximum tolerated dose of GCSF in mobilizing circulating CD34+ hematopoietic stem cells, with the limiting dose based on GCSF-related severe adverse effects. A one-month safety of GCSF will be tested with the 2 standard doses of 5 ug/kg/d and 10 ug/kg/d.

ELIGIBILITY:
Inclusion Criteria:

1. Completed the preliminary work up for cholestasis with suspected or inconclusive diagnosis of BA
2. Gestational Age > 36wks
3. Weight > 2 Kg
4. Age >-2 weeks-<180 days at diagnosis
5. Serum Direct Bilirubin > 2 mg/dL GGT > 100 U/L
6. Kasai operated patients for Type 3 or 4 anatomy of BA
7. Cholangiogram/porta hepatis findings diagnostic of BA
8. Liver biopsy supporting BA diagnosis

Exclusion Criteria:

1. Having access to liver transplantation for immediate Kasai failure
2. Prior Kasai patients
3. Major cardiac, renal, CNS malformations with poor prognosis
4. Intracranial hemorrhage
5. History of recent TPN use within the last 2 weeks of surgery
6. GI tract obstruction
7. Laparoscopic Kasai repair

Ages: 2 Weeks to 180 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Dose determination GCSF | 13 months
  To determine the maximum tolerated dose of GCSF based on GCSF dose limiting toxicity and the extent of peripheral blood stem cell mobilization as measured by increases in CD34+cells with upper levels limited by white blood cells (WBCs) less than 50,000 per microliter (mcL) of blood.

CONTACTS AND LOCATIONS:
Overall Officials: Evan P Nadler, MD, Principal Investigator — Children's National Research Institute
Locations (2):
- Children's National Medical Center, Washington D.C., District of Columbia, United States
- National Childrens Hospital, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Davenport M. Biliary atresia: clinical aspects. Semin Pediatr Surg. 2012 Aug;21(3):175-84. doi: 10.1053/j.sempedsurg.2012.05.010. PMID 22800970
- [Background] Panopoulos AD, Watowich SS. Granulocyte colony-stimulating factor: molecular mechanisms of action during steady state and 'emergency' hematopoiesis. Cytokine. 2008 Jun;42(3):277-88. doi: 10.1016/j.cyto.2008.03.002. Epub 2008 Apr 8. PMID 18400509
- [Background] Yannaki E, Athanasiou E, Xagorari A, Constantinou V, Batsis I, Kaloyannidis P, Proya E, Anagnostopoulos A, Fassas A. G-CSF-primed hematopoietic stem cells or G-CSF per se accelerate recovery and improve survival after liver injury, predominantly by promoting endogenous repair programs. Exp Hematol. 2005 Jan;33(1):108-19. doi: 10.1016/j.exphem.2004.09.005. PMID 15661404
- [Background] Takami T, Terai S, Sakaida I. Stem cell therapy in chronic liver disease. Curr Opin Gastroenterol. 2012 May;28(3):203-8. doi: 10.1097/MOG.0b013e3283521d6a. PMID 22395569
- [Background] Prajapati R, Arora A, Sharma P, Bansal N, Singla V, Kumar A. Granulocyte colony-stimulating factor improves survival of patients with decompensated cirrhosis: a randomized-controlled trial. Eur J Gastroenterol Hepatol. 2017 Apr;29(4):448-455. doi: 10.1097/MEG.0000000000000801. PMID 27930386
- [Derived] Nguyen HPA, Ren J, Butler M, Li H, Qazi S, Sadiq K, Dao HT, Holterman A. Study protocol of Phase 2 open-label multicenter randomized controlled trial for granulocyte-colony stimulating factor (GCSF) in post-Kasai Type 3 biliary atresia. Pediatr Surg Int. 2022 Jul;38(7):1019-1030. doi: 10.1007/s00383-022-05115-0. Epub 2022 Apr 7. PMID 35391541